CLINICAL TRIAL: NCT02177799
Title: Surveillance Study of Acute Gastroenteritis in Hospitalized Children
Brief Title: Surveillance Study of Acute Gastroenteritis in Hospitalized Children in Rural Area in Lebanon
Acronym: SAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaikh Ragheb Harb Hospital (Other)
Responsible Party: Principal Investigator, HADI FAKIH, MD, Hadi FAKIH MD, Shaikh Ragheb Harb Hospital
Other Study IDs: RHH12014
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Acute Gastroenteritis; Diarrhea; Rotavirus
Keywords: Gastroenteritis; Hospitalized; Children
MeSH Terms: conditions — Diarrhea; Gastroenteritis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gastroenteritis

SUMMARY:
Acute gastroenteritis is a common cause of hospitalization in children with significant socioeconomic burden on the health community, we will follow in this observational and analytical study the admitted cases of acute gastroenteritis to the pediatric floor at the Sheikh Ragheb Harb Hospital over a period of summer time to determine the causes, etiologies and epidemiology of Age in a community hospital.

DETAILED DESCRIPTION:
In this survey of hospitalized cases of acute gastroenteritis, children between two months and up to ten years old are included except for known cases of chronic diarrhea, malnutrition or immunodeficiency, data collected include clinical signs and symptoms, epidemiologic information and laboratory data during the hospital stay, also hospital treatment will be reviewed to determine the therapeutic options available in our country and its convenience with the disease and clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* children with acute gastroenteritis admitted to the pediatric floor

Exclusion Criteria:

* chronic diarrhea or Immunodeficiency

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children male and female from 2 months to 10 year old
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Age distribution | one year after completing data collection

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Ragheb Harb Hospital, Nabatieh, Toul, Lebanon